CLINICAL TRIAL: NCT03306212
Title: Effectiveness of Intermittent Serial Casting on Spastic Wrist Flexion Deformity in Children With Cerebral Palsy Treated By Botulinum Toxin A
Brief Title: Efficacy of Intermittent Serial Casting on Spastic Wrist Flexion Deformity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nigar Dursun, Head of PMR Department, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KOU KAEK 2014/269
Record Dates: First submitted 2017-10-05; First posted 2017-10-10 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; casting; Botulinum toxin A
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA; Occupational Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Casting Group (Experimental): Patients treated by botulinum toxin A and occupational therapy and intermittent serial casting
  Interventions: Drug: Botulinum toxin A; Other: Occupational Therapy; Other: Intermittent serial casting
- Control Group (Active Comparator): Patients treated by botulinum toxin A and occupational therapy
  Interventions: Drug: Botulinum toxin A; Other: Occupational Therapy

INTERVENTIONS:
Drug: Botulinum toxin A
  Other Names: Dysport
Other: Occupational Therapy
Other: Intermittent serial casting
  Arms: Casting Group

SUMMARY:
Spastic wrist flexion deformity is a very common problem in children with CP. Although serial casting (SC) is one of the commonly used interventions in addition to botulinum toxin A (BoNT-A) injections and physical therapy for spastic deformities of lower extremity of children with CP, there is limited data on SC in the upper extremity.

In this prospective, randomized, controlled clinical trial in order to overcome the issues with patient compliance, side effects and combined treatment options an intermittent SC model was developed. The objective of this study was to show the effects of intermittent SC when combined with occupational therapy (OT) and BoNT-A injections on spasticity, and passive range of motion (pROM) of children with CP having spastic wrist flexion deformity.

DETAILED DESCRIPTION:
Spasticity is not only the most common motor disorder but also the main cause of slowly developing secondary problems like contractures in children with cerebral palsy (CP). Spastic wrist flexion deformity is a very common problem in children with CP and can be primarily due to spasticity of the palmar muscle complex, can be exacerbated by the weakness of the antagonist dorsiflexor muscles and can involve soft tissue and joint contractures. Although serial casting (SC) is one of the commonly used interventions in addition to botulinum toxin A (BoNT-A) injections and physical therapy for spastic deformities of lower extremity of children with CP, there is limited data on SC in the upper extremity. Skin irritation or breakdown, painful epizodes, oedema, tendonitis, weakness, stiffness are some of the side effects reported after SC. Moreover casting especially when prolonged might complicate activities of daily living for instance by increasing the risk of falls or causing problems in bathing. Recent evidence from literature favors early, goal oriented, activity based, intensive, repetitive motor trainings in enriched environments to optimize neuroplasticity in children with CP. Prolonged serial casting might also interfere with these activity based, intensive rehabilitation options for upper extremity.

In this prospective, randomized, controlled clinical trial in order to overcome the issues with patient compliance, side effects and combined treatment options an intermittent SC model was developed. The objective of this study was to show the effects of intermittent SC when combined with occupational therapy (OT) and BoNT-A injections on spasticity, and passive range of motion (pROM) of children with CP having spastic wrist flexion deformity.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis of CP according to Rosenbaum criteria,
* having a unilateral spastic palmar flexion deformity of wrist joint,
* having a Modified Ashworth Scale (MAS) score of 3 in the palmar flexor muscle complex,
* being scheduled for BoNT-A treatment to upper extremity including palmar flexor muscle group.

Exclusion Criteria:

* having cognitive dysfunction,
* having a history of orthopedic surgery to upper extremity,
* having significant dystonia,
* having infection skin breakdown,
* having vascular disease,
* having fracture or dislocation.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline Passive ROM | 12 weeks
  Range of motion measurement
Mean change from baseline MAS score | 12 weeks
  Tone measurement

SECONDARY OUTCOMES:
Mean change from XV3 angle of Tardieu scale | 12 weeks
  Spasticity measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No